CLINICAL TRIAL: NCT02228785
Title: Study of the Safety and Tolerance of Three Doses of G17DT in Patients With Metastatic Colorectal Cancer.
Brief Title: A Study of the Safety and Tolerance of Three Doses of G17DT in Metastatic Colorectal Cancer
Acronym: CC1C
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor local tolerance to injection.
Sponsor: Cancer Advances Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CC1C
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 100µg dose of G17DT (Experimental): Patients in this arm received a 100µg dose of G17DT via intramuscular injection.
  Interventions: Biological: G17DT
- 200µg dose of G17DT (Experimental): Patients in this arm received a 200 µg dose of G17DT via intramuscular injection.
  Interventions: Biological: G17DT
- 500µg dose of G17DT (Experimental): Patients in this arm received a 500µg dose of G17DT via intramuscular injection.
  Interventions: Biological: G17DT

INTERVENTIONS:
Biological: G17DT
  Other Names: Polyclonal Antibody Stimulator

SUMMARY:
This study was designed to investigate the safety and tolerance of three doses (100µg, 200µg, 500µg) of G17DT for the treatment of patients with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or over with histologically verified adenocarcinoma of colon or rectum.
* Recurrent of metastatic disease not amenable to curative surgery and/or radiotherapy.
* Life expectancy greater than 3 months.
* Karnofsky Index Score greater than or equal to 50%.
* Written informed consent obtained.

Exclusion Criteria:

* Neoplastic lesions other than colorectal cancer (except treated basal cell carcinoma of the skin or cancer of the uterine cervix, through Stage I.
* Acute intercurrent illness.
* Patient considered to be a medical risk because of non-malignant systemic disease or grossly abnormal laboratory results.
* Patients who had received any other anticancer therapy within 3 months.
* Factor liable to alter the serum gastrin concentration or affect intra-gastric acidity, for instance concomitant therapy with H2 receptor antagonist drugs, proton pump inhibitors, or previous gastric surgery.
* Patients immunologically compromised including those on corticosteroid therapy.
* Women of child-bearing age.
* Positive immediate hypersensitivity reaction to skin testing with study medication.
* Patients unable to complete the diary book
* Haematogical Status Haemoglobin count less than 10g/dL White Blood Cell count less than 4.0 x 10^9/L Platelet count less than 100 x 10^9/L

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1994-05; Primary Completion 1994-10 (Actual)

PRIMARY OUTCOMES:
Injection Site Reaction | Through Week 12
  An examination was performed to assess injection site tolerability at every posttreatment visit.
Antibody Levels | Through Week 12
  Gastrin-17 antibodies are produced as a result of treatment with G17DT and the proportion of patients producing gastrin-17 antibodies was considered to be an appropriate measure of the immunogenicity of the dosing schedule under study.

SECONDARY OUTCOMES:
Intra-gastric pH | Through Week 8
  Compare the pre-immunization 24-hour intra-gastric pH with post-immunization profiles.

CONTACTS AND LOCATIONS:
Overall Officials: J D Hardcastle, MChir, FRCP, FRCS, Principal Investigator — University of Nottingham